CLINICAL TRIAL: NCT03723122
Title: Cancer-related Communication Between Patients and Their Caregivers: A Randomized Controlled Trial Assessing the Efficacy of a Dyadic Communication Reinforcement Intervention (DCRI)
Brief Title: Efficacy of a Dyadic Cancer-related Communication Reinforcement Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Darius Razavi, Prof., Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DCRI
Record Dates: First submitted 2018-10-23; First posted 2018-10-29 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Cancer; Communication Programs
Keywords: Psychological intervention; Dyadic communication; Dyadic adaptation to cancer
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization allocation is given only at the data manager. Participant, care provider and assessor do not know in which group participants are allocated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCRI program (Experimental): Patient-caregiver dyads will immediately attend the Dyadic communication reinforcement intervention. For both groups, first assessment time take place just after the enrollment, before the randomization. For this group, second assessment time take place 2 weeks post-intervention. Pre-post assessments consist in self-reported scales assessing emotional distress, individual coping, cancer-related dyadic communication frequency, satisfaction, self-efficacy and coping.
  Interventions: Behavioral: Dyadic Communication Reinforcement Intervention
- Waiting List (No Intervention): Patient-caregiver dyads are in a waiting condition for 6 weeks. They will attend the Intervention after the second assessment time if they want to. For both group, first assessment time take place just after the enrollment, before the randomization. For this group, second assessment time take place 6 weeks after first assessment time. First and second assessment consist in self-reported scales assessing emotional distress, individual coping, cancer-related dyadic communication frequency, satisfaction, self-efficacy and coping.

INTERVENTIONS:
Behavioral: Dyadic Communication Reinforcement Intervention — Psycho-educative and behavioral intervention centered on cancer-related dyadic communication
  Arms: DCRI program

SUMMARY:
Background: To face cancer-related stress, patients and caregivers activate individual and dyadic coping responses. Opened communication, adequate involvement, reciprocal supportive roles, self-disclosure and responsiveness enhance dyadic coping. Nevertheless, little is known about the optimal content of dyadic interventions designed to improve dyadic communication.

Methods: A randomized controlled trail was designed to assess the efficacy of a dyadic intervention centered on a cancer-related communication reinforcement. Patient-caregiver dyads are randomly assigned to either an intervention group or a waiting list group. Patients and caregivers complete self-reported scales that assessed emotional distress, individual coping, cancer-related dyadic communication frequency, satisfaction, self-efficacy and coping at baseline and post-treatment (intervention group), or 6 weeks after baseline (waiting list group). This dyadic communication reinforcement intervention (DCRI) consists of a weekly 4-session intervention. This intervention includes specific communication tasks aiming the improvement of some cancer-related dyadic communication competencies such as concerns disclosure and request for support.

Discussion: DCRI would lead to improvements in cancer-related dyadic communication self-efficacy, cancer-related dyadic communication satisfaction and dyadic coping.

DETAILED DESCRIPTION:
1. Aim of the trial: A randomized longitudinal study assessing the efficacy of a dyadic communication reinforcement intervention (DCRI) between cancer patients and their caregivers. Efficacy of the DCRI will be assessed by the analysis of changes over time in both patients and caregivers self-reported questionnaires/scales measures.
2. Participants: Patients and caregivers are recruited from oncology clinics at Erasme Hospital and Jules Bordet Institute (Brussels, Belgium). Recruitment and all study procedures were approved by a central ethics committee (Erasme - ULB Ethics Committee) and all participants are providing written informed consent.
3. Study Design: Participants are randomly assigned to the experimental group, consisting of the DCRI, or to the control group, consisting of a waiting list. Dyads in the waiting list can complete the DCRI after the last assessment if they want to. Investigator, psychologist in charge of the intervention and participants are blinded for this randomization. Dyads completed a follow-up assessment (T2), either 2 weeks after the DCRI in the experimental group or 6 weeks after baseline in the control condition. All assessment time were completed either at the outpatient clinic or at home.
4. DCRI content: DCRI aims communication reinforcement by a weekly 4-sessions program. DCRI is manualized and is conducted by an experienced psychologist (same psychologist for all participating dyads). Sessions focus on reciprocal cancer-related stress communication between patients and their caregivers using a specific communication task that promotes self-disclosure and request for support. All sessions are divided into four times: (1) session introduction, (2) first communication task, (3) second communication task and (4) session conclusion.

(1)Session introduction: Firstly, psychologist assesses if any significant moment occurred before the actual session and let dyad members talk about it if they want. Secondly, psychologist addresses some theoretical information about the session subject. First and second session subject is about personal cancer-concerns disclosure and close one supportive response to this disclosure. Third and fourth session subject is about personal request for support to face a cancer-related stress and close one response to this request for support. In the first and second session, psychologist therefore discusses the importance of sharing stress appraisal, stress describing, thoughts and emotions expressing and how to be supportive in responding. In the third and fourth session, psychologist discusses the importance of the personal needs communication and the clarity of the request for support to be well understood by the partner.

(2 & 3) First and second communication task: This communication task is divided into an audio-recorded communication exercise and the debriefing of this communication exercise. In each session, there are therefore two communication tasks (two exercises and two debriefing). An exercise lasts 5 minutes and psychologist stays with the dyad but does not intervene during it. This exercise consists in patient and caregivers embody a specific role: "discloser" and "listener". Each role is associated with specific instructions. Exercise (and therefore task) is performed twice a session to let patient and caregiver experiment each of these roles. In the first and second session, the discloser has to express a personal cancer-related stress to the listener. The listener has to listen and respond supportively to this expressed cancer-related stress. In the third and fourth session, the discloser has to ask for help about a personal cancer-related stress to the listener. The listener has to listen and respond to this request for support. The exercise debriefing consists in the listening, in session, of the exercise record. After the listening, psychologist asks to the listener what kind of the discloser communicational behavior help him to understand the expressed cancer-related stress. Psychologist asks also to the discloser what kind of the listener communicational behavior help him to feel supported. After that, psychologist reinforces each positive communication strategy used by the discloser and the listener.

(4) Session conclusion: Psychologist summarizes the two communication tasks and notes all positive communication strategies used by the patient and the caregiver in self-disclosing/responding (first and second session) or request for support/responding to request for support.

5. Assessment procedure: Patients and caregivers are assessed by self-reported measures at baseline (T1) (after enrollment) and 2 weeks after the intervention (in the experimental group) or 6 weeks after baseline (T2) (in the control group). Patients and caregivers complete exactly the same self-reported questionnaires and scales. Patients had a medical information questionnaire in addition at baseline and study personnel rated their performance status, based on the Karnofsky Performance Status Scale, at T1 and T2. Other specific oncologic information was collected by medical record review.

At T1, demographic questionnaire assesses gender, age, cultural background, education level, native speaking, professional situation, familial situation (children) and psychiatric history. At T1, dyadic information questionnaire assesses relationship type, relationship length, living situation and contact frequency between patients and caregivers.

Patients and caregivers complete following self-reported scales in T1 and T2: (1) Cancer-related dyadic communication frequency, (2) cancer-related dyadic communication satisfaction, (3) cancer-related communication self-efficacy, (4) Dyadic Coping Inventory, (5) Hospital Anxiety and Depression Scale and (6) Ways of Coping Checklist.

6. Statistical Analysis: Statistical analysis consisted in a comparative analysis of groups at baseline using parametric and nonparametric tests as appropriate (Student's t test, Mann-Withney U test or Chi-squared test). Patients and caregivers outcomes at baseline and after the DCRI, or after the waiting period, were compared using repeated measures analysis of variance (MANOVA). Time and group-by-time effects were processed using MANOVA. Effect size will be report with eta-squared (η²) given by MANOVA. All tests were two-tailed, and the alpha was set at 0.05. All analyzes were performed using SPSS®, version 25.

7. Data Quality Control: There are 6 study collaborators: (1) recruitment manager, (2) investigation coordinator, (3) assessor, (4) psychologist in charge of the intervention, (5) data manager and (6 & 7) two data assistants.

1. Recruitment manager manages the recruitment process. Every recruitment steps have been approved by institution ethics committee. Patients phone numbers meeting inclusion criteria are provided by the medical staff to the recruitment manager only. These phone numbers are destroyed after the recruitment phase. Recruitment manager calls each patient to give them basic information about the study. If they are interested in, recruitment manager calls the designated caregiver with the patient consent. If the caregiver agrees too, recruitment manager makes an appointment to provide a written informed consent.
2. Investigation assistant provides the randomization number for each participating dyad to the data manager. He books all DCRI session for the psychologist in the good time lapses (regarding the group).
3. Assessor assists participants in questionnaires and scales if they need it and he rates each patient by a Karnofsky score. A numerical copy is made for each assessment. This copy is put on a encrypted hard drive disk. Paper version is given in person to data manager. Paper versions are stored in a secure location.
4. Psychologist conducts the DCRI
5. Data manager manages randomization number, securing data storage, data encoding and encoding checking.
6. Data assistants encode data provide by the questionnaires and scales. They only have a participant ID and no randomization information. Double encoding, checked by the data manager, reduces encoding error.

This 7-persons functioning guarantees complete masking procedure from recruitment to encoding.

ELIGIBILITY:
Inclusion Criteria:

* To read and speak French
* To be aged 18 years old or more
* To be diagnosed with any cancer type with a life expectancy of ≥ 6 months or be the caregiver of patients meeting this inclusion criteria
* To benefit from a folfox, folfiri, folfirinox or folfiri+bevacizumab-type chemotherapy with a life expectancy of ≥ 6 months or be the caregiver of patients meeting this inclusion criteria

Exclusion Criteria:

* Not be treated for a psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Cancer-related dyadic communication | 2 months
  Cancer-related dyadic communication self-efficacy through a self-reported scale for patients and caregivers. The perceived dyadic communication self-efficacy was measured by a 6-dimension scale: Dyadic Communication Competencies. Each dimension is divided into 5 items. Subject has to rate each item on a 0-100 range (0 = not certain; 100 = absolutely certain) to report how he is certain to matser the communication competency. A total score (ranging 0-100) for each dimension is computed by making the mean of all item scores. A higher score reflects a higher perceived communication self-efficacy.
Dyadic coping | 2 months
  Cancer-related dyadic coping through a validated self-reported scale for patients and caregivers: Dyadic Coping Inventory (DCI). It is composed of the following six different dimensions: stress communication, supportive dyadic coping, delegated dyadic coping, negative dyadic coping, common dyadic coping and evaluation of dyadic coping. The DCI has a 5-point Likert scale (1 = "Rarely"; 5 = "Very Frequently") and provides a total score (35-175) by summing all items. A higher score reflects a better dyadic coping.

SECONDARY OUTCOMES:
Emotional Distress | 2 months
  Emotional distress levels through a validated self-reported scale for patients and caregivers: The Hospital Anxiety and Depression Scale (HADS). It is composed by 2 dimensions (anxiety and depression) and has a 4-point Likert scale that vary at each item. HADS provides a total score (0-42 range) by summing all item scores. A higher score reflects a higher emotional distress. Anxiety subscale score (0-21 range) is providen by summing all Anxiety-items. A higher score reflects more anxiety. Depression subscale scores (0-21 range) is providen by summing all Depression-items. A higher score reflects more depression.

CONTACTS AND LOCATIONS:
Overall Officials: Darius Razavi, MD, PhD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Hopital Erasme & Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
The plan is under review

REFERENCES:
- [Background] Lee E, Roberts LJ. (2018). Between individual and family coping: a decade of theory and research on couples coping with health-related stress. Journal of Family Theory & Review 10: 141-164. doi: 10.1111/jftr.12252.
- [Background] Kayser K, Watson LE, Andrade JT. (2007). Cancer as a "We-disease": examining the process of coping from a relational perspective. Family Systems & Health 25(4): 404-418.
- [Background] Candy B, Jones L, Drake R, Leurent B, King M. Interventions for supporting informal caregivers of patients in the terminal phase of a disease. Cochrane Database Syst Rev. 2011 Jun 15;(6):CD007617. doi: 10.1002/14651858.CD007617.pub2. PMID 21678368
- [Background] Li Q, Loke AY. A literature review on the mutual impact of the spousal caregiver-cancer patients dyads: 'communication', 'reciprocal influence', and 'caregiver-patient congruence'. Eur J Oncol Nurs. 2014 Feb;18(1):58-65. doi: 10.1016/j.ejon.2013.09.003. Epub 2013 Oct 4. PMID 24100089
- [Background] Song L, Rini C, Ellis KR, Northouse LL. Appraisals, perceived dyadic communication, and quality of life over time among couples coping with prostate cancer. Support Care Cancer. 2016 Sep;24(9):3757-65. doi: 10.1007/s00520-016-3188-0. Epub 2016 Apr 2. PMID 27039207
- [Background] Badr H, Krebs P. A systematic review and meta-analysis of psychosocial interventions for couples coping with cancer. Psychooncology. 2013 Aug;22(8):1688-704. doi: 10.1002/pon.3200. Epub 2012 Oct 9. PMID 23045191
- [Background] Waldron EA, Janke EA, Bechtel CF, Ramirez M, Cohen A. A systematic review of psychosocial interventions to improve cancer caregiver quality of life. Psychooncology. 2013 Jun;22(6):1200-7. doi: 10.1002/pon.3118. Epub 2012 Jun 25. PMID 22729992
- [Background] Manne SL, Ostroff JS, Norton TR, Fox K, Goldstein L, Grana G. Cancer-related relationship communication in couples coping with early stage breast cancer. Psychooncology. 2006 Mar;15(3):234-47. doi: 10.1002/pon.941. PMID 15926198
- [Background] Northouse LL, Mood DW, Montie JE, Sandler HM, Forman JD, Hussain M, Pienta KJ, Smith DC, Sanda MG, Kershaw T. Living with prostate cancer: patients' and spouses' psychosocial status and quality of life. J Clin Oncol. 2007 Sep 20;25(27):4171-7. doi: 10.1200/JCO.2006.09.6503. Epub 2007 Jul 16. PMID 17635953
- [Background] Kayser K, Scott J. (2008). Helping couples cope with women's cancer. New York : Springer.
- [Background] Manne S, Badr H, Zaider T, Nelson C, Kissane D. Cancer-related communication, relationship intimacy, and psychological distress among couples coping with localized prostate cancer. J Cancer Surviv. 2010 Mar;4(1):74-85. doi: 10.1007/s11764-009-0109-y. Epub 2009 Dec 6. PMID 19967408
- [Background] Porter LS, Keefe FJ, Baucom DH, Hurwitz H, Moser B, Patterson E, Kim HJ. Partner-assisted emotional disclosure for patients with gastrointestinal cancer: results from a randomized controlled trial. Cancer. 2009 Sep 15;115(18 Suppl):4326-38. doi: 10.1002/cncr.24578. PMID 19731357
- [Background] Porter LS, Keefe FJ, Baucom DH, Hurwitz H, Moser B, Patterson E, Kim HJ. Partner-assisted emotional disclosure for patients with GI cancer: 8-week follow-up and processes associated with change. Support Care Cancer. 2012 Aug;20(8):1755-62. doi: 10.1007/s00520-011-1272-z. Epub 2011 Sep 24. PMID 21947440
- [Derived] Tiete J, Delvaux N, Lienard A, Razavi D. Efficacy of a dyadic intervention to improve communication between patients with cancer and their caregivers: A randomized pilot trial. Patient Educ Couns. 2021 Mar;104(3):563-570. doi: 10.1016/j.pec.2020.08.024. Epub 2020 Aug 27. PMID 33129628